CLINICAL TRIAL: NCT02379312
Title: Comparison of the Satiety Effect of a Very Low Energy Foam With Normal Energy Foams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-NAA-0291
Record Dates: First submitted 2015-02-17; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-01

CONDITIONS: Satiety; Appetite
Keywords: Foams; Satiety; Appetite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Very low energy aerated beverage (Active Comparator): Very low energy aerated beverage
  Interventions: Dietary Supplement: Very low energy aerated beverage
- Normal energy aerated beverage 1 (Active Comparator): Normal energy aerated beverage 1
  Interventions: Dietary Supplement: Normal energy aerated beverage 1
- Normal energy aerated beverage 2 (Active Comparator): Normal energy aerated beverage 2
  Interventions: Dietary Supplement: Normal energy aerated beverage 2
- Normal energy aerated beverage 3 (Active Comparator): Normal energy aerated beverage 3
  Interventions: Dietary Supplement: Normal energy aerated beverage 3

INTERVENTIONS:
Dietary Supplement: Very low energy aerated beverage
  Arms: Very low energy aerated beverage
Dietary Supplement: Normal energy aerated beverage 1
  Arms: Normal energy aerated beverage 1
Dietary Supplement: Normal energy aerated beverage 2
  Arms: Normal energy aerated beverage 2
Dietary Supplement: Normal energy aerated beverage 3
  Arms: Normal energy aerated beverage 3

SUMMARY:
To compare, in a randomized, single-blinded, cross-over study the satiety effect of a very low energy aerated beverage with normal energy aerated beverages in healthy subjects.

DETAILED DESCRIPTION:
The primary objective of this study is to assess if a very low energy foam has the same effect on satiety as the same volume of a reference normal energy foam, by testing for equivalence of these two foams. Treatment equivalence, is met if the 90% confidence interval (CI) of between-treatment differences in appetite AUC is within the range of -5 to +5 mm/min of the reference . Two other normal energy foams with slightly different compositions are also compared to the reference foam to test for possible effects of differences in composition (carbohydrate type, emulsifier) other than energy per se.

On each test day, volunteers will arrive at the clinic in a fasted state where they consume a standardized 250 kcal breakfast. Subjects receive one of the four test products 2.5 hours after start of breakfast and consume 400 ml of the test products with a spoon within 10 minutes. Each subject will be randomized to a treatment order according to a balanced (Williams type) design, and receive one of four test products each week for 4 weeks, separated by a one-week washout period (consumed on the same week day).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 30 kg/m² (inclusive)
* Apparently healthy: no medical conditions which might effect study measurements (judged by study physician).

Exclusion Criteria:

* Dislike, allergy or intolerance to test products
* Eating disorder (measured by SCOFF questionnaire, > 2 "yes" responses)
* High or very high restrained eater measured by Three factor eating questionnaire TFEQ, restriction score > 14
* Reported medical treatment that may affect eating habits/satiety

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Hunger and satiety questions | Time points -155, -90, -5, 15, 30, 60, 90, 120, 150 and 180 min
  Area under the time curve of hunger and satiety scores (as rated by the subjects on a Visual Analog Scale)

SECONDARY OUTCOMES:
Electronic Visual Analogue Scale (EVAS) for liking questions | Time point 15 min

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Blanc, PhD, Study Director — Eurofins Optimed